CLINICAL TRIAL: NCT01505075
Title: Phase II Study of Dose-escalated, Hypofractionated Radiotherapy and Androgen Deprivation Therapy for High-Risk Prostate Cancer
Brief Title: Safety and Efficacy Study of Hypofractionated Radiotherapy and Androgen Deprivation Therapy for Prostate Cancer
Acronym: pHART8
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Sunnybrook Health Sciences Centre (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 043-2011
Record Dates: First submitted 2011-10-05; First posted 2012-01-06 (Estimated); Last update posted 2020-11-24 (Actual); Status verified 2020-11

CONDITIONS: Prostate Cancer
Keywords: prostatic neoplasms; radiotherapy; hypofractionated; high risk prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Radiation Dose Hypofractionation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Hypofractionated radiation (Experimental): 40 Gy in 5 fractions over 29 to prostate; 30 Gy in 5 fractions over 29 days to seminal vesicles
  Interventions: Radiation: Hypofractionated radiation

INTERVENTIONS:
Radiation: Hypofractionated radiation — 40 Gy in 5 fractions to prostate, 30 Gy in 5 fractions to seminal vesicles; total treatment duration 29 days
  Other Names: RapidArc

SUMMARY:
The purpose of this study is to determine the safety and efficacy of a short course of radiotherapy (40Gy/5 fractions/29 days) for the treatment of high risk prostate cancer currently being managed with primary androgen deprivation therapy (PADT).

DETAILED DESCRIPTION:
Primary Endpoints:

* Acute gastrointestinal (GI) and genitourinary (GU) Common Terminology Criteria for Adverse Events (CTCAE) v3.0 toxicities

Secondary Endpoints:

* Late GI and GU Radiation Therapy Oncology Group (RTOG) toxicities
* Biochemical disease-free survival
* Biopsy positive rate at 3 years
* Quality of life using the Expanded Prostate Cancer Index Composite (EPIC) questionnaire
* Develop a biobank of DNA and serum extracted from blood and urine to analyze and develop new biomarkers for prostate cancer progression or susceptibility to severe toxicity

ELIGIBILITY:
Inclusion Criteria:

* informed consent obtained
* men > 18 years
* histologically confirmed prostate adenocarcinoma (centrally reviewed)
* high risk prostate cancer, defined as at least one of: clinical stage T3, or gleason score 8-10, or PSA > 20ng/mL

Exclusion Criteria:

* prior pelvic radiotherapy
* anticoagulation medication (if unsafe to discontinue for gold seed insertion)
* diagnosis of bleeding diathesis
* pelvic girth > 40cm (to ensure visibility of gold seeds on electronic portal imaging)
* large prostate (> 90cm3) on imaging
* severe lower urinary tract symptoms (International Prostate Symptom Score >19 or nocturia > 3)
* No evidence of castrate resistance (defined as PSA < 3ng/mL while testosterone is < 0.7nmol/L). Patients could have been on combined androgen blockade but are excluded if this was started due to PSA progression

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2011-09 (Actual); Primary Completion 2013-01 (Actual); Study Completion 2021-09 (Estimated)

PRIMARY OUTCOMES:
Incidence of grade 3+ rectal toxicity | Acute period (up to 3 months)
  Common Terminology Criteria for Adverse Events (CTCAE) v3.0

SECONDARY OUTCOMES:
Incidence of grade 3+ urinary toxicity | Acute (up to 3 months) and Late (after 6 months of follow-up)
  Common Terminology Criteria for Adverse Events (CTCAE) v3.0
Quality of Life | 5 years
  Expanded Prostate Cancer Index Composite (EPIC)
Biochemical (ie.prostate specific antigen) disease free survival | 5 years
Incidence of grade 3+ rectal toxicity | Late (after 6 months of follow-up)
  Common Terminology Criteria for Adverse Events (CTCAE) v3.0

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Loblaw, MD, FRCPC, Principal Investigator — Sunnybrook Health Sciences Centre; Suneil Jain, MD, Principal Investigator — suneil.jain@sunnybrook.ca
Locations (1):
- Odette Cancer Centre, Sunnybrook Health Sciences Centre, Toronto, Ontario, Canada